CLINICAL TRIAL: NCT06997094
Title: Phase I Decitabine Dose-Tolerance in Surgically Resectable HPV-Negative Head and Neck Cancer
Brief Title: Decitabine in Combination With Standard of Care Therapy for the Treatment of Surgically Resectable HPV-Negative Head and Neck Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC240706; NCI-2025-03537 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-012507 (Other: Mayo Clinic Institutional Review Board); MC240706 (Other: Mayo Clinic)
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Human Papillomavirus-Negative Neck Squamous Cell Carcinoma; Resectable Head and Neck Squamous Cell Carcinoma; Resectable Human Papillomavirus-Independent Head and Neck Mucosal Squamous Cell Carcinoma; HPV-Negative Squamous Cell Carcinoma; Resectable Head and Neck Squamous-cell Carcinoma
MeSH Terms: interventions — Specimen Handling; Drug Therapy; Decitabine; Injections; Congresses as Topic; Radiation; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (decitabine, surgery, radiation) (Experimental): PREOPERATIVE PHASE: Patients receive decitabine IV over 1 hour QD for 3 days and undergo standard of care surgery within 28 days of receiving decitabine.
  ADJUVANT TREATMENT: Patients receive decitabine IV over 1 hour QD for 3 days every 3 weeks during radiation therapy in the absence of disease progression or unacceptable toxicity. Patients also undergo EBRT QD on 5 days per week for up to 5-35 treatments per standard of care. Patients may receive concurrent chemotherapy of choice per standard of care.
  Patients also undergo blood sample collection throughout the study.
  Interventions: Procedure: Biospecimen Collection; Drug: Chemotherapy; Drug: Decitabine; Radiation: External Beam Radiation Therapy; Other: Questionnaire Administration; Procedure: Surgical Procedure

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Chemotherapy — Given concurrent chemotherapy
  Other Names: Chemo; Chemotherapy (NOS); Chemotherapy, Cancer, General
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2'-deoxycytidine; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Radiation: External Beam Radiation Therapy — Undergo EBRT
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam Radiotherapy (conventional); External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam; Teleradiotherapy; Teletherapy; Teletherapy Radiation
Other: Questionnaire Administration — Ancillary studies
Procedure: Surgical Procedure — Undergo standard of care surgery
  Other Names: Operation; Surgery; Surgery Type; Surgery, NOS; Surgical; Surgical Intervention; Surgical Interventions; Surgical Procedures; Type of Surgery

SUMMARY:
This phase I trial tests the safety, side effects, and best dose of decitabine in combination with standard of care surgery, radiation, and/or chemotherapy and the effectiveness of the combination in treating patients with head and neck squamous cell cancers that are not caused by human papilloma virus (HPV-negative) and that can be removed by surgery (resectable). Decitabine, an antimetabolite, stops cells from making deoxyribonucleic acid (DNA) and may kill tumor cells. Studies have shown that medications like decitabine can make some types of solid tumors more sensitive to chemotherapy. This allows the chemotherapy to be more effective, with slower progression and longer survival. Decitabine is also a clinically active demethylating agent, and may help make tumor cells more sensitive to radiation therapy. Radiation therapy uses high energy x-rays, particles, or radioactive seeds to kill tumor cells and shrink tumors. External beam radiation therapy (EBRT) is a type of radiation that uses a machine to aim high-energy rays at the tumor from outside the body. Chemotherapy drugs work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving decitabine in combination with standard of care surgery, radiation and/or chemotherapy may be safe, tolerable, and/or effective in treating patients with surgically resectable HPV-negative head and neck squamous cell cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To prospectively evaluate the maximum tolerated dose (MTD) of decitabine, in both the preoperative and adjuvant phases of treatment, combined with standard-of-care therapy including surgery +/- chemoradiation for HPV-negative head and neck cancers.

SECONDARY OBJECTIVES:

I. Evaluation of acute (early onset) toxicities. (Stratified by methylation status) II. Evaluation of late onset toxicities. (Stratified by methylation status) III. Evaluation of event-free survival (EFS). (Stratified by methylation status) IV. Evaluation of overall survival (OS). (Stratified by methylation status) V. Evaluation of quality of life (QOL). (Stratified by methylation status)

CORRELATIVE RESEARCH OBJECTIVES:

I. In vivo methylation response to preoperative decitabine. II. Pharmacokinetics of decitabine. III. Exploratory circulating biomarkers.

OUTLINE: This is a dose-escalation study followed by a dose-expansion study.

PREOPERATIVE PHASE: Patients receive decitabine intravenously (IV) over 1 hour once daily (QD) for 3 days and undergo standard of care surgery within 28 days of receiving decitabine.

ADJUVANT TREATMENT: Patients receive decitabine IV over 1 hour QD for 3 days every 3 weeks during radiation therapy in the absence of disease progression or unacceptable toxicity. Patients also undergo EBRT QD on 5 days per week for up to 5-35 treatments per standard of care. Patients may receive concurrent chemotherapy of choice per standard of care.

Patients also undergo blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 30 days, every 4-6 months for 2 years and then every 12 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* REGISTRATION: Age ≥ 18 years
* REGISTRATION: Histologic confirmation of HPV-negative, squamous cell carcinoma of the head and neck that is surgically resectable. HPV-status confirmation by p16, circulating tumor DNA or in-situ hybridization is only required for oropharyngeal primaries

  * Includes mucosal and non-mucosal subsites
  * Includes head and neck of unknown primary origin REGISTRATION: Measurable disease preoperatively, as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or equivalent criteria
  * NOTE: Tumor lesions in a previously irradiated area are not considered measurable disease; disease that is measurable by physical examination only is not eligible
* REGISTRATION: Absence of distant metastases on standard diagnostic work-up ≤ 16 weeks prior to registration. (chest computed tomography [CT] or positron emission tomography [PET]/CT)
* REGISTRATION: Negative pregnancy test done ≤ 7 days prior to registration, for women of childbearing potential only

  * NOTE: If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* REGISTRATION: Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* REGISTRATION: Hemoglobin ≤ 9.0 g/dL (obtained ≤ 14 days prior to registration)
* REGISTRATION: Absolute neutrophil count (ANC) ≥ 1500/mm^3 (obtained ≤ 14 days prior to registration)
* REGISTRATION: Platelet count ≥ 100,000/mm^3 (obtained ≤ 14 days prior to registration)
* REGISTRATION: Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (obtained ≤ 14 days prior to registration)
* REGISTRATION: Alanine aminotransferase (ALT) and aspartate transaminase (AST) ≤ 3 x ULN (≤ 5 x ULN for patients with liver involvement) (obtained ≤ 14 days prior to registration)
* REGISTRATION: Prothrombin time (PT)/international normalized ratio (INR)/activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN (obtained ≤ 14 days prior to registration) OR if patient is receiving anticoagulant therapy and INR or aPTT is within target range of therapy
* REGISTRATION: Provide written informed consent
* REGISTRATION: Ability to complete questionnaire(s) by themselves or with assistance
* REGISTRATION: Willingness to provide mandatory blood specimens for correlative research
* REGISTRATION: Willingness to provide mandatory tissue specimens for correlative research
* REGISTRATION: Willing to return to enrolling institution for follow-up (during the active monitoring phase of the study)
* RE-REGISTRATION FOR ADJUVANT DOSE ASSIGNMENT: Patient received pre-operative decitabine dose
* RE-REGISTRATION FOR ADJUVANT DOSE ASSIGNMENT: The patient had study-specific surgery
* RE-REGISTRATION FOR ADJUVANT DOSE ASSIGNMENT: Patient meets adjuvant radiation criteria based on investigator choice

Exclusion Criteria:

* REGISTRATION: Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women who are of childbearing potential who are unwilling to employ adequate contraception
* REGISTRATION: Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* REGISTRATION: Immunocompromised patients and patients known to be HIV positive and currently receiving antiretroviral therapy

  * NOTE: Patients known to be HIV positive, but without clinical evidence of an immunocompromised state, are eligible for this trial
* REGISTRATION: Failure to recover from acute, reversible effects of prior therapy regardless of interval since last treatment

  * EXCEPTION: Grade 1 peripheral (sensory) neuropathy that has been stable for at least 3 months since completion of prior treatment
* REGISTRATION: Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Or psychiatric illness/social situations that would limit compliance with study requirements
* Dyspnea at rest due to complications of advanced malignancy or other disease that requires continuous oxygen therapy
* REGISTRATION: Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* REGISTRATION: Other active malignancy ≤ 5 years prior to registration

  * EXCEPTIONS: Non-melanotic skin cancer or carcinoma-in-situ of the cervix
  * NOTE: If there is a history of prior malignancy, they must not be receiving other specific treatment for their cancer
* REGISTRATION: History of myocardial infarction ≤ 6 months, or congestive heart failure requiring use of ongoing maintenance therapy for life-threatening ventricular arrhythmias
* REGISTRATION: Prior history of radiation therapy to the affected site
* REGISTRATION: Prior systemic chemotherapy ≤ 5 years prior to registration for other diagnosis not related to study disease
* REGISTRATION: Contraindication to radiation therapy as determined by the treating team
* REGISTRATION: Contraindication to decitabine as determined by the treating team
* RE-REGISTRATION FOR ADJUVANT DOSE ASSIGNMENT: Experienced a dose limiting toxicity (DLT) during pre-operative decitabine therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-23 (Actual); Primary Completion 2027-11-08 (Estimated); Study Completion 2027-11-08 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of preoperative decitabine | From first dose of preoperative decitabine to the first dose of adjuvant decitabine
  MTD will be selected based on the rate of grade 4 toxicity and correlative methylation response data.
MTD of adjuvant decitabine | From first dose of adjuvant decitabine to 28 days after the end of treatment
  MTD will be selected based on the rate of grade 4 toxicity and correlative methylation response data.

SECONDARY OUTCOMES:
Incidence of acute (early onset) adverse events | Up to 90 days
  Defined as toxicities which begin during the start of adjuvant therapy until 90 days post end of treatment. Will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The maximum grade for each type of acute AE will be recorded for each patient.
Incidence of late onset adverse events | From 91 days to 2 years
  Defined as toxicities which begin from 91 days to two years post radiation therapy. Early onset toxicities can also be considered late toxicities if they persist for at least one day beyond the 90 days used to define late onset toxicities. Will be assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The maximum grade for each type of acute AE will be recorded for each patient.
Event-free survival | 1 year, 2 years, 5 years
  Defined as the interval from registration to last follow-up without an event, defined to include 1) recurrence of disease, 2) progression of disease, or 3) death.
Overall survival | 1 year, 2 years, 5 years
  Defined as the interval from registration to last follow-up or death from any cause.
Quality of Life - EORTC QLQ-H&N35 | Baseline, at end of treatment, every 4-6 months post end of treatment for up to 2 years
  Assessed using the EORTC (European Organization for Research and Treatment of Cancer) QLQ (Quality of Life) - Head & Neck 35 (H&N35) inventory, a 35-item questionnaire that assesses symptoms encountered specifically by patients with head and neck cancer. This measure generates 7 multiple-item scales (Pain, Swallowing, Senses, Speech, Social eating, Social contact, and Sexuality), in addition to 11 single items (e.g., opening mouth, sticky saliva, dry mouth). Scales range in score from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning whereas a high score for a symptom scale or item represents a high level of symptomatology or problems.

CONTACTS AND LOCATIONS:
Overall Officials: Adam L. Holtzman, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials